CLINICAL TRIAL: NCT03258242
Title: A Randomized, Double-masked, Multicenter, Placebo Controlled Study of Keluo Xin Capsule on Efficacy and Safety in Patients With Diabetic Retinopathy
Brief Title: A Study of Keluo Xin Capsule Compare to Placebo in Terms of Efficacy and Safety in Patients With Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Kanghong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH105-B02-CRP-2.0
Record Dates: First submitted 2017-08-04; First posted 2017-08-23 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Moderately Severe to Severe NPDR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Keluo Xin Capsule (Experimental)
  Interventions: Drug: Keluo Xin capsule
- Placebo Comparator: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Keluo Xin capsule — four capsules at a time, three times a day, taken orally and consecutively for 24 weeks or 48 weeks.
  Arms: Experimental: Keluo Xin Capsule
Drug: Placebo oral capsule — four placebo capsules at a time, three times a day, taken orally and consecutively for 24 weeks or 48 weeks.
  Arms: Placebo Comparator: Placebo

SUMMARY:
This is a study aiming to assess the efficacy and safety of Keluo Xin capsule in patients with moderately severe to severe nonproliferative diabetic retinopathy (NPDR). Two-thirds of participates will receive Keluo Xin capsules while other one third will receive placebo.

DETAILED DESCRIPTION:
This study composes two parts. The first is a 24-week period during which subjects receive designed treatment regimen; after that, subjects will be informed again for the next 24-week regimen (extention phase) and can choose whether or not to participate in the treatment (with the same regimen in the first period) voluntarily.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 70 years;
* Patients diagnosed with type 2 diabetes mellitus;
* Patients diagnosed with nonproliferative diabetic retinopathy;
* Patients diagnosed with traditional Chinese medicine syndrome(TCM) differentiation of both Qi and Yin deficiency with blood Stasis;
* HbA1c≤8.0%;

Exclusion Criteria:

* Study eye been received panretinal photocoagulation;
* Study eye with neovascular elsewhere or neovascular of the disc, or neovascularization of iris;
* Prior panretinal photocoagulation in the study eye within 6 months;
* Uncontrolled blood pressure;
* Subjects who develop chronic diarrhoea;
* Any history of acute diabetic complications;
* Any history of allergy to components of Keluo Xin capsule;
* Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-08-31 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change from DR severity as measured by the early treatment diabetic retinopathy score chart at 24 weeks | Baseline and 24 weeks
  Based on the classification criteria of Early Treatment of Diabetic Retinopathy Study to grade DR severity.
Mean change from DR severity as measured by the early treatment diabetic retinopathy score chart at 48 weeks | Baseline and 48 weeks
  Based on the classification criteria of Early Treatment of Diabetic Retinopathy Study to grade DR severity.
Pathological changes from baseline at 24 weeks as measured by optical coherence tomography (OCT) . | Baseline and 24 weeks
Pathological changes from baseline at 48 weeks as measured by optical coherence tomography (OCT) . | Baseline and 48 weeks
Pathological changes from baseline at 24 weeks as measured by fluorescence angiography (FFA). | Baseline and 24 weeks
Pathological changes from baseline at 48 weeks as measured by fluorescence angiography (FFA). | Baseline and 48 weeks
Mean change from baseline in Chinese medicine syndrome score chart at 24 weeks | Baseline and 24 weeks
  The score chart is based on the typical symptoms and signs both in the eye and whole body on patients with DR and is used to assess DR severity.
Mean change from baseline in Chinese medicine syndrome score chart at 48 weeks | Baseline and 48 weeks
  The score chart is based on the typical symptoms and signs both in the eye and whole body on patients with DR and is used to assess DR severity.

SECONDARY OUTCOMES:
Mean change from baseline in best corrected visual acuity at 24 weeks | Baseline and 24 weeks
  Visual acuity is assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Mean change from baseline in best corrected visual acuity at 48 weeks | Baseline and 48 weeks
  Visual acuity is assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Frequency and severity of ocular and non-ocular adverse events over time | Screening to 24 weeks and 48 weeks

OTHER OUTCOMES:
Change of retinal blood flow density | Baseline and 24 weeks
  A exploratory objective which will be evaluated by angio OCT.
Change of retinal blood flow density | Baseline and 48 weeks
  A exploratory objective which will be evaluated by angio OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Song, Professor, Principal Investigator — Wuhan General Hospital of Guangzhou Military, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Academy of Ophthalmology, "Diabetic retinopathy.," 2014.
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281